CLINICAL TRIAL: NCT06632314
Title: Impact of Enteral Feeding on Cerebral and Splanchnic Oxygenation During Packed Red Blood Cell Transfusion in Preterm Infants: a Prospective Randomized Controlled Study
Brief Title: Impact of Enteral Feeding on Splanchnic Oxygenation During Packed Red Blood Cell Transfusion in Preterm Infants
Acronym: TANEC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Hakan Ongun, Associate professor in neonatology, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: KAEK-737
Record Dates: First submitted 2024-10-07; First posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Necrotizing Enterocolitis of Newborn; Feeding Intolerance; PreTerm Neonate; Transfusion Related Complications
Keywords: enteral feeding; splanchnic oxygenation; preterm neonate; transfusion related necrotizing enterocolitis; NIRS
MeSH Terms: interventions — Enteral Nutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Feeding continued arm (Active Comparator): Enteral feeding will continue during packed red blood cell transfusion. Regional cerebral and splanchnic oxygenation will be measured using near-infrared spectroscopy (NIRS) for 48 hours. Cerebral and splanchnic oxygenation parameters, including cerebral regional oxygen saturation (crSO2), splanchnic regional oxygen saturation (srSO2), the ratio of crSO2 to srSO2 (CSOR), cerebral fractionated tissue oxygen saturation (cFTOE) and splanchnic fractionated tissue oxygen saturation (sFTOE) will be measured immediately before PRBCT (baseline) and at the first, sixth, 12th, 24th, and 48th hours after PRBCT using near-infrared spectroscopy.
  Interventions: Dietary Supplement: Enteral feeding
- Feeding restricted arm (Active Comparator): Enteral feeding will be withhold during packed red blood cell transfusion. Regional cerebral and splanchnic oxygenation will be measured using near-infrared spectroscopy (NIRS) for 48 hours. Cerebral and splanchnic oxygenation parameters, including cerebral regional oxygen saturation (crSO2), splanchnic regional oxygen saturation (srSO2), the ratio of crSO2 to srSO2 (CSOR), cerebral fractionated tissue oxygen saturation (cFTOE) and splanchnic fractionated tissue oxygen saturation (sFTOE) will be measured immediately before PRBCT (baseline) and at the first, sixth, 12th, 24th, and 48th hours after PRBCT using near-infrared spectroscopy.
  Interventions: Dietary Supplement: Enteral feeding

INTERVENTIONS:
Dietary Supplement: Enteral feeding — Enteral feeding will be withheld or continued in very low birthweight neonates during packed red blood cell transfusion. Regional cerebral and splanchnic oxygenation will be measured using near-infrared spectroscopy (NIRS) for 48 hours. Cerebral and splanchnic oxygenation parameters, including cerebral regional oxygen saturation (crSO2), splanchnic regional oxygen saturation (srSO2), the ratio of crSO2 to srSO2 (CSOR), cerebral fractionated tissue oxygen saturation (cFTOE) and splanchnic fractionated tissue oxygen saturation (sFTOE) will be measured immediately before PRBCT (baseline) and at the first, sixth, 12th, 24th, and 48th hours after PRBCT using near-infrared spectroscopy.
  Other Names: enteral nutrition

SUMMARY:
This clinical trial aims to learn if enteral feeding influences cerebral and splanchnic oxygenation during red blood cell infusion in very low birth-weight preterm infants. It will also learn about how continuing or withholding enteral feeding during blood transfusion might trigger transfusion-related necrotizing enterocolitis. The main questions, it aims to answer are:

* Does continuing or withholding enteral feeding have any impact on splanchnic and cerebral oxygenation in very-low-birth-weight preterm infants?
* Does continuing enteral feeding result in feeding intolerance during red blood cell infusion or transfusion-related necrotizing enterocolitis (TANEC) in very-low-birth-weight preterm infants? Researchers will compare regional cerebral and splanchnic oxygenation obtained by Near Infra-Red Spectroscopy (NIRS) monitoring while receiving red blood cell transfusion.

Participants will:

* Continue or withhold enteral feeding during red blood cell infusion, and all participants will be under NIRS monitoring for the following 48 hours after the blood transfusion.
* Be monitored for any signs and symptoms of new-onset feeding intolerance and/or necrotizing enterocolitis for 48 hours following the blood transfusion

DETAILED DESCRIPTION:
Continuing enteral feeding during red blood cell transfusion can have a negative impact on cerebral and splanchnic oxygenation and trigger transfusion-related necrotizing enterocolitis (TANEC) in very low birth-weight infants of gestational age less than 32 weeks and/or birthweight less than 1500 grams. However, the issue of continuing or withholding enteral feeding to prevent TANEC in these neonates is a matter of debate. Enteral feeding is often withheld during blood transfusion to prevent TANEC.

This study was carried out to investigate the effect of enteral feeding during red blood cell infusion on cerebral and splanchnic oxygenation in low-birth-weight preterm infants. Secondary hypothesis was to observe (if any) the signs and symptoms of a new-onset feeding intolerance and/or necrotizing enterocolitis for 48 hours following the blood transfusion.

Enteral feeding will continue or be withhold in very low birthweight neonates during packed red blood cell transfusion. Regional cerebral and splanchnic oxygenation were measured using near-infrared spectroscopy (NIRS) for 48 hours.

ELIGIBILITY:
Inclusion Criteria:

1. infants with gestational age ≤32 weeks and/or birthweight ≤1500 gr,
2. survival at least the first week of life
3. being able to tolerate a minimum total daily feeding volume of 100 mL/kg/day,
4. hemodynamically stable infant (no need of inotropic support)
5. receiving packed red blood cell transfusion for the treatment of anemia of prematurity

Exclusion criteria:

1. feeding intolerance
2. newly or previously diagnosed stage II and greater necrotizing enterocolitis
3. spontaneous intestinal perforation
4. suspected / proven sepsis in the previous 72 hours
5. neonates in need of high-frequency oscillated ventilation support,
6. previous PRBC transfusions due to iatrogenic anemia, hemolysis and/or intraventricular hemorrhage to avoid sensitization by blood products,
7. hemodynamically significant patent ductus arteriosus
8. history of abdominal surgery,
9. complex congenital anomalies involving gastrointestinal tract and cardiovascular system,
10. missing data,
11. parental reluctance to consent.

Ages: 1 Day to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Splanchnic oxygenation | Prior to red blood cell transfusion to 48 hours following blood transfusion
  Monitoring regional splanchnic oxygenation (SrSO2) and splanchnic fractionated tissue oxygen saturation (sFTOE)
Cerebral oxygenation | Prior to red blood cell transfusion to 48 hours following blood transfusion
  Monitoring Cerebral oxygenation parameters, including cerebral regional oxygen saturation (crSO2), cerebral fractionated tissue oxygen saturation (cFTOE)

SECONDARY OUTCOMES:
Feeding intolerance and/or transfusion related necrotizing enterocolitis | Prior to red blood cell transfusion to 48 hours following blood transfusion
  To observe (if any) the signs and symptoms of a new-onset feeding intolerance and/or necrotizing enterocolitis for next 48 hours following the blood transfusion.

CONTACTS AND LOCATIONS:
Overall Officials: Hakan ONGUN, MD, Principal Investigator — Akdeniz university faculty of medicine department of pediatrics, division of neonatology
Locations (1):
- Akdeniz University Faculty of Medicine, Antalya, Konyaalti, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Patient data (excluding patient name, ID and parental consent forms) will be shared
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: November 2024 - November 2025
Access Criteria: The datasets generated during and/or analysed during the current study will be available upon request from Hakan ONGUN